CLINICAL TRIAL: NCT04351165
Title: An Open-Label, Randomized, Single-Dose, 2-Way Crossover Study to Compare the Bioavailability of Two IMP4297 Formulations (20 mg Capsules and 10 mg Capsules) After Single Oral Administration of 100 mg IMP4297 Under Fasted Condition in Healthy Male Subjects
Brief Title: BA Study of IMP4297 (20mg vs 10mg) in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Impact Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IMP4297-107
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Solid Tumor
MeSH Terms: interventions — senaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Period 1:
  100 mg oral dose of IMP4297 (5 capsules, 20 mg/capsule);
  Period 2:
  100 mg oral dose of IMP4297 (10 capsules, 10 mg/capsule);
  Each treatment sequence will consist of 2 periods, separated by a washout period of at least 7 days between each Dose.
  Interventions: Drug: IMP4297
- Arm 2 (Experimental): Period 1:
  100 mg oral dose of IMP4297 (10 capsules, 10 mg/capsule);
  Period 2:
  100 mg oral dose of IMP4297 (5 capsules, 20 mg/capsule);
  Each treatment sequence will consist of 2 periods, separated by a washout period of at least 7 days between each Dose.
  Interventions: Drug: IMP4297

INTERVENTIONS:
Drug: IMP4297 — IMP4297 10mg/capsule; IMP4297 20mg/capsule;

SUMMARY:
An open-label, randomized, single-dose, 2-way crossover study to compare the bioavailability of two IMP4297 formulations (20 mg capsules and 10 mg capsules) after single oral administration of 100 mg IMP4297 under fasted condition in healthy male subjects

DETAILED DESCRIPTION:
This will be an open-label, randomized, single-dose, 2-way crossover study to compare the bioavailability of two IMP4297 formulations (10 mg capsules and 20 mg capsules) after single oral administration of 100 mg IMP4297 under fasted condition in healthy male subjects. It will be conducted at one site, and approximately a total of 18 subjects will be enrolled.

Subjects will be randomized to one of the 2 treatment sequences according to a computer-generated randomization schedule. Each treatment sequence will consist of 2 periods, separated by a washout period of at least 7 days between each period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects, 18 to 55 years of age (both inclusive) on the day of signing informed consent form (ICF).
2. Body Mass Index (BMI) of 18 to 30 kg/m2 (both inclusive); and a total body weight 50 kg.
3. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, physical examination, including blood pressure (BP), pulse rate (PR) measurement, temperature, 12-lead ECG, or clinical laboratory tests, etc., judged by the investigator. For example, the reference normal ranges (inclusive) are as follows: after at least 5-minute rest in a supine position, BP: 90-139/60-89 mmHg, and PR: 50-100 bpm. Repeat assessment can be conducted at the discretion of the investigator or delegate.
4. Subjects able to father children must use a highly effective non-drug contraception double barrier method for the duration of the study and for at least 90 days after the last dose of study medication and should not have any plan for sperm donation throughout this period. Note: Sexual abstinence is allowed if this is the preferred and usual lifestyle of the subject. Male subjects are also eligible to participate if they have a bilateral vasectomy or have a female partner of non-childbearing potential.
5. Subjects must voluntarily participate in this study. Be willing and be able to provide written informed consent for this clinical trial. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
6. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Evidence or history of clinically significant diseases, including but not limited to neurologic, cardiovascular, hematological, immunological, renal, hepatic, gastrointestinal, pulmonary, endocrine, metabolic, psychiatric, or allergic disease (including drug and food allergies).
2. Any condition possibly affecting drug absorption (e.g., gastrectomy, difficulty in swallowing).
3. General anesthesia within 3 months before administration, or have a planned surgery during the study period.
4. History of drug abuse within the past 5 years, or a positive urine drug test at screening or the admission. Repeat assessment can be conducted at the discretion of the investigator or delegate.
5. History of excessive alcohol intake exceeding 10 drinks/week (1 standard drink = 150 mL of wine, 360 mL of beer, or 45 mL of hard liquor) within 3 months prior to screening, or a positive alcohol breath test at screening or the admission. Repeat assessment can be conducted at the discretion of the investigator or delegate.
6. Use of tobacco or nicotine containing products in excess of the equivalent of 5 cigarettes per day within 3 months prior to screening, a positive urine nicotine test at screening or the admission, or difficulty abstaining from smoking for the duration of study confinement. Repeat assessment can be conducted at the discretion of the investigator or delegate.
7. Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to the first dose of study drug; participation in a clinical trial of device(s) within 30 days prior to the first dose of study drug; participation in ≥4 clinical trials within one year prior to the first dose of study drug.
8. Blood donation (excluding plasma donations) or significant loss of blood (≥400 mL) within 1 month prior to screening, received blood transfusion or use of blood products.
9. Use of any medicinal product that changes the activity of hepatic enzymes within 28 days prior to the first dose of study drug, such as potent CYP3A4 inhibitors or inducers, or subjects who need to continue receiving these medications during the study period (refer to Appendix 18.2 for the list of common CYP3A4 inhibitors or inducers).
10. Use of prescription or nonprescription drugs, dietary supplements, or herbal medicines, within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study drug. As an exception, paracetamol may be used at doses of ≤1 g/day. Limited use of nonprescription medications that are not believed to affect the overall results of the study may be permitted on a case by case basis following approval by the principal investigator and the sponsor.
11. Subjects with history of hepatitis, or positive result at screening for hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), hepatitis C antibody (HCVAb), or human immunodeficiency virus antibody (HIVAb).
12. Screening supine 12-lead ECG demonstrating a QTcF (using Fridericia's formula, QTcF = QT/RR1/3) interval >450 msec, or a QRS interval >120 msec. If QTcF >450 msec or QRS >120 msec, the ECG should be repeated 2 more times and the average of the 3 QTcF or QRS values should be used to determine the subject's eligibility.
13. Unable to abstain from strenuous exercise within 48 hours prior to dosing and during the study period.
14. Use of products containing alcohol, tobacco, nicotine, caffeine within 48 hours prior to dosing; or unable to abstain from using these products for the duration of study confinement.
15. History of sensitivity to any ingredients of IMP4297 products evaluated in this study.
16. History of hemophobia, inability to tolerate venipuncture, and being afraid of needles.
17. Subjects who have received live vaccine within 28 days prior to screening.
18. Any other medical or psychiatric condition that may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for study participation.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Cmax | 3 months
  peak concentration
AUC0-last | 3 months
  area under the curve from time zero to the time with the last quantifiable concentration
AUC0-inf | 3 months
  area under the curve from time zero to infinity

SECONDARY OUTCOMES:
Safety endpoints | 3 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.03
Tmax | 3 months
  time to reach Cmax
t½ | 3 months
  elimination half-life
CL/F | 3 months
  apparent clearance
Vz/F | 3 months
  apparent volume of distribution

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Health, Sydney, Australia

IPD SHARING:
Plan to Share IPD: Undecided